CLINICAL TRIAL: NCT03831529
Title: Prognostic Factors Associated With Mortality Within 6 Months Among Critically Ill Elderly Patients Admitted to the Intensive Care Unit With Severe Acute Cholangitis
Brief Title: Outcomes of Elderly Patients Admitted to the Intensive Care Unit With Severe Acute Cholangitis
Acronym: ANGIOCHOLREA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/ANGIOCHOLREA-NOVY/NK
Record Dates: First submitted 2019-01-18; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Cholangitis Infective; Elderly Person
Keywords: critically ill; mortality; outcome; treatment intensity level
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU older patient: Older patient (> 65 years old) admitted to ICU with severe acute cholangitis

SUMMARY:
The aging of the population goes along with an increased demand for intensive care among very elderly patients (above 75-80 years old). At the same time, there is a decline in the supply of intensive care units (ICU). The 1-year mortality of patients above 80 years old in ICU ranged from 40 to 70%. Moreover, many survivors suffer from long-term sequelae as poor quality of life, cognitive impairment and functional disability.

It is unclear under what conditions older patients may benefit from ICU admission. Cholangitis frequently occured in older patient. Moreover, severe acute cholangitis is a potentially life threatening disease characterized by a biliary obstruction and an infection of the bile possibly evolving towards systemic infection, shock and death. Because of its potential rapid reversibility of symptom thanks to early intravenous antibiotics and biliary decompression with drainage, old patients suffering from acute cholangitis are easily admitted to intensive care unit.

To date, there is a lack of data about the outcome in this population admitted to the intensive care unit with acute cholangitis.

The aim of the current study is to describe the outcomes in elderly patients (> 75 years old) admitted to the ICU with acute cholangitis and to identify prognostics factors associated with long term mortality (6 months).

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* ICU admission for acute cholangitis
* follow up in the same center after the ICU stay

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients > 65 years old admitted to the ICU for acute severe cholangitis
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
mortality | 180 days
  rate of survivors and non survivors

SECONDARY OUTCOMES:
mortality | 90 days
  rate of survivors and non survivors
mortality | 28 days
  rate of survivors and non survivors
factors associated with 6 months mortality (underlying condition) | Day 1
  Functional status : presence or absence of denutrition defined by a BMI < 19 kg/m2 and/or albuminemia < 30 g/l and/or loss of weight > 5% during the last month (or > 10% during the last three months)
factors associated with 6 months mortality (severity score) | Day 1
  Simplified Acute Physiology Score 2 Minimum value : 0 / Maximun value 163
factors associated with 6 months mortality (Presence of hemodynamic failure) | Up to 7 days
  infusion of catecholamine (ie norepinephrine) during the ICU stay, yes or not
factors associated with 6 months mortality (Presence of respiratory failure) | Up to 7 days
  number of day(s) under mechanical ventilation
factors associated with 6 months mortality (Presence of renal failure) | Up to 7 days
  number od day(s) under renal replacement therapy
Clinical evolution | Day 3
  Change in Sequential Organ Failure score between Day 1 and Day 3. We measured the Sepsis-related Organ Failure Assessment (SOFA) score at day and day 3 and then made the difference between the two scores the SOFA score could range between 0 and 24 We calculated the score at day 1 and day 3 and made the difference An absence or a small difference between the 2 days is associated with a worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHR Mercy, Metz, Lorraine
  - Emmanuel NOVY, Vandœuvre-lès-Nancy, Lorraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novy E, Carrara L, Remen T, Chevaux JB, Losser MR, Louis G, Guerci P. Prognostic factors associated with six month mortality of critically ill elderly patients admitted to the intensive care unit with severe acute cholangitis. HPB (Oxford). 2021 Mar;23(3):459-467. doi: 10.1016/j.hpb.2020.08.003. Epub 2020 Aug 22. PMID 32839088